CLINICAL TRIAL: NCT03174886
Title: A 24-month Randomised Parallel Group Single-blinded Multi-centre Phase 1 Pilot Study of AADvac1 in Patients With Non Fluent Primary Progressive Aphasia
Brief Title: A 24-month Phase 1 Pilot Study of AADvac1 in Patients With Non Fluent Primary Progressive Aphasia
Acronym: AIDA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Axon Neuroscience SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-TP-001; 2017-000643-41 (EudraCT Number)
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Primary Progressive Nonfluent Aphasia
Keywords: tau; neurofibrillary; degeneration; primary progressive aphasia; agrammatic; tauopathy; immunotherapy; immunization
MeSH Terms: conditions — Primary Progressive Nonfluent Aphasia; Pick Disease of the Brain; Aphasia, Primary Progressive; Tauopathies | interventions — AADvac1

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to one of two dosage strengths of AADvac1. No placebo is used. No active comparator is used.
Who Masked: Participant
Masking Description: Patients are unaware of the dosage strength they are receiving. The AADvac1 vials are numbered, and the coding unknown to the patient. The investigator handles the vaccine vials and administers the IMP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AADvac1 40 µg (Experimental): The intervention consists of Axon Peptide 108 coupled to keyhole limpet haemocyanin (KLH) 40 µg/0.30 mL suspension for injection; and aluminium hydroxide Al(OH)3 (containing approx. 0.5 mg Al3+/0.30 mL), administered subcutaneously. The basic immunisation regimen consists of 6 doses administered subcutaneously in 6-week intervals. Subsequently, 5 booster doses are applied in 13-week intervals, for a total of 11 administrations.
  Interventions: Drug: AADvac1 40 µg
- AADvac1 160 µg (Experimental): The intervention consists of Axon Peptide 108 coupled to KLH 160 µg/0.30 mL suspension for injection; and aluminium hydroxide Al(OH)3 (containing approx. 0.5 mg Al3+/0.30 mL), administered subcutaneously. The basic immunisation regimen consists of 6 doses administered subcutaneously in 6-week intervals. Subsequently, 5 booster doses are applied in 13-week intervals, for a total of 11 administrations.
  Interventions: Drug: AADvac1 160 µg

INTERVENTIONS:
Drug: AADvac1 40 µg — Active immunotherapy against neurofibrillary pathology.
  Arms: AADvac1 40 µg
Drug: AADvac1 160 µg — Active immunotherapy against neurofibrillary pathology.
  Arms: AADvac1 160 µg

SUMMARY:
This study is a pilot trial evaluating the safety and immunogenicity of AADvac1 in patients with the non-fluent variant of Primary Progressive Aphasia.

50% of participants will receive the 40 µg dosage of AADvac1 and 50% of participants will receive the 160 µg dosage of AADvac1. No placebo is used.

DETAILED DESCRIPTION:
The non-fluent variant of Primary progressive Aphasia (nfvPPA) is a chronic progressive neurodegenerative disorder of the brain. Over the course of the disease, pathological proteins accumulate in the brain, damaging neurons, thus causing them to lose their connections and die.

No treatments are currently available; symptomatic medications are used off-label in nfvPPA.

AADvac1 is designed to raise antibodies against pathological tau protein (the primary constituent of neurofibrillary pathology, which is the underlying cause of disease in ~80% of nfvPPA cases). These antibodies are expected to prevent tau protein from aggregating, to facilitate the removal of tau protein aggregates and prevent the spreading of pathology, slowing or halting the progress of the disease.

ELIGIBILITY:
Inclusion criteria

1. Patient has a clinical diagnosis of non-fluent/agrammatic variant PPA according to the criteria by Gorno-Tempini et al. (2011) with evidence of left frontal brain hypometabolism. Patients with right-sided hypometabolism are eligible for the study only if they are left-handed.
2. Patient has a FTLD-CDR language domain score of ≤ 2, and other individual FTLD-CDR domain scores ≤ 1.
3. Patient's age is 18 - 85 years inclusive at the time of having provided informed consent.
4. Patient has adequate visual and auditory abilities and premorbid local language skills to allow neuropsychological testing.
5. Sexually active female patients must be using highly effective contraception methods, or be surgically sterile, or be at least 2 years post-menopausal.
6. Sexually active male patients must be using highly effective contraception methods, or be surgically sterile.
7. Patient and caregiver have signed and dated written informed consent.
8. Availability of a partner/caregiver knowing the patient and being able to accompany the patient to the visits.
9. Patient is legally competent.

Exclusion Criteria:

1. The patient's brain MRI is incompatible with a diagnosis of nfvPPA.
2. Patient has a history or evidence of a central nervous system (CNS) disorder other than nfvPPA which may cause symptoms of aphasia or dementia (Alzheimer's disease, Dementia with Lewy Bodies, inflammatory/demyelinating CNS conditions, Creutzfeldt-Jakob disease, Huntington's disease, etc.)
3. Patient has a history or currently suffers from a significant psychiatric illness such as schizophrenia, any type of psychotic disorder or bipolar affective disorder.
4. Patient has a history or evidence of cerebrovascular disease (ischemic or haemorrhagic stroke), or diagnosis of possible, probable or definite vascular dementia.
5. Patient has Wernicke's encephalopathy.
6. Patient has metabolic or toxic encephalopathy or dementia due to a general medical condition.
7. Patient suffers from hypothyroidism, defined as thyroid-stimulating hormone elevation > 5.000 mcIU/mL, and/or fT4 levels < 0.7 ng/dL. Patients with corrected hypothyroidism are eligible for the study provided that treatment has been stable for 12 weeks before study entry.
8. Patient has a known pathogenic mutation in GRN or C9orf72.
9. Presence or history of allergy to components of the vaccine.
10. Presence and/or history of immunodeficiency (e.g., HIV).
11. Patient is currently being treated with immunosuppressive drugs.
12. Patient has a history and/or currently suffers from a clinically significant autoimmune disease, or is expected to receive immunosuppressive or immunomodulatory treatment at the present or in the future.
13. Patient has a recent (≤ 5 years since last specific treatment) history of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia).
14. Patient has an active infectious disease (e.g., Hepatitis B, C).
15. Patient had a myocardial infarction within the last 2 years.
16. Patient has a current clinically important systemic illness that is likely to result in deterioration of the patient's condition or affect the subject's safety during the study:

    1. poorly controlled congestive heart failure (New York Heart Association [NYHA] score ≥ 3),
    2. poorly controlled diabetes,
    3. severe renal insufficiency (Estimated glomerular filtration rate < 30 mL/min),
    4. chronic liver disease - ALT (alanine aminotransferase) > 2x upper limit of normal range (ULN), AST (aspartate aminotransferase) > 2x ULN
    5. other clinically significant systemic illness, if considered relevant by the investigator.
17. Patient had alcohol or drug dependence within the past year.
18. Patient has a current diagnosis of epilepsy.
19. Pregnant or breastfeeding women.
20. Patient has participated in another interventional clinical trial within 12 weeks before Visit 01.
21. Patient has contraindication for MRI imaging such as metallic endoprosthesis or MRI-incompatible stent implantation.
22. Patient has contraindications for other study procedures, such as CSF sampling.
23. Patient had surgery (under general anaesthesia) within 12 weeks prior to Visit 01 and/or scheduled surgery (under general anaesthesia) during the whole study period.
24. Patient is currently being treated or was treated in the past with any active vaccines for a neurodegenerative disorder.
25. Patients not expected to complete the clinical trial.
26. Patient, in the opinion of the investigator, is unlikely to comply with the clinical study protocol, or is unsuitable for other reasons.
27. Patient is dependent from Sponsor or investigator (e.g. as an employee or as a relative).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 25 months
  The safety assessment is based on the number, type and severity of adverse events (AEs).
Immunogenicity (Percentage of patients who develop an IgG immune response, geometric mean titre of titre of antibodies against Axon Peptide 108, IgG to IgM ratio of antibodies against Axon Peptide 108) | 24 months
  AADvac1 depends on raising antibodies that mediate its treatment effects. Immunogenicity assessment includes: Percentage of AADvac1-treated patients who develop an immune response (responder rate), geometric mean titre of antibodies against Axon Peptide 108, IgG to IgM ratio of antibodies against Axon Peptide 108.

OTHER OUTCOMES:
Cerebrospinal fluid (CSF) biomarkers | 24 months
  Temporal change in total CSF neurogranin, phosphorylated neurofilament heavy chain protein, ubiquitin, β-synuclein, tau protein, phospho-tau pT181, N-terminal tau protein, amyloid β1-40, amyloid-β1-42, ubiquitin, α-, β- and γ-synuclein, Chitinase-3-like protein (YKL-40), Monocyte chemoattractant protein-1 (MCP-1), and other CSF markers
Serum neurofilament light chain protein (and other blood biomarkers of nfvPPA) | 24 months
  Temporal change in neurofilament light chain protein and other blood biomarkers (exploratory measure; biomarker panel to be finalised based on the state of the art at the time of analysis)
Magnetic resonance imaging (MRI) volumetry | 24 months
  Temporal change in whole brain volume and set of regions of interest, as measured by MRI
Frontotemporal lobar degeneration - Clinical Dementia Rating - Sum of Boxes (FTLD-CDR-SB) | 24 months
  Temporal change in FTLD-CDR SB score
Clinician's Global Impression - Improvement (CGI-I) | 24 months
  Temporal change in CGI-I score
Instrumental Activities of Daily Living (IADL) | 24 months
  Temporal change in Amsterdam IADL
Custom Cognitive Battery | 24 months
  Temporal change in the custom Cognitive Battery score
Addenbrooke's Cognitive Examination | 24 months
  Temporal change in Addenbrooke's Cognitive Examination score
Unified Parkinson's disease rating scale (UPDRS) part III | 24 months
  Temporal change in UPDRS part III score
Frontal Systems Behavior Scale (FrSBe) | 24 months
  Temporal change in FrSBe score
Immune cell (granulocyte, monocyte, and lymphocyte populations) | 24 months
  Temporal change in immunological variables (monocytes, lymphocytes, basophil and neutrophil granulocytes; a range of lymphocyte sub-populations - CD3+, CD3+/CD4+, CD3+/CD4+/CD28+, CD3+/CD4+/CD28+/CD45RA+, CD3+/CD4+/CD28+/CD45RO+, CD3+/CD8+, CD3+/CD8+/CD28+, CD3+/CD8+/CD28+/CD45RA+, CD3+/CD8+/CD28+/CD45RO+) over 24 months
Correlation of a range of potential immunological predictors with IgG antibody titres against Axon Peptide 108 | 24 months
  Correlation of measures of immune response with immunological variables (monocytes, lymphocytes, basophil and neutrophil granulocytes; a range of lymphocyte sub-populations - CD3+, CD3+/CD4+, CD3+/CD4+/CD28+, CD3+/CD4+/CD28+/CD45RA+, CD3+/CD4+/CD28+/CD45RO+, CD3+/CD8+, CD3+/CD8+/CD28+, CD3+/CD8+/CD28+/CD45RA+, CD3+/CD8+/CD28+/CD45RO+) will individually be assessed for correlation with IgG antibody titres. The possibility of multiple independent predictors of the antibody response will be examined using regression trees analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Otto, Prof, Principal Investigator — Universitat Ulm
Locations (3):
- Germany (3):
  - Universitätsmedizin Göttingen, Klinik für Psychiatrie und Psychotherapie, Göttingen
  - Klinikum Rechts der Isar der TU München, Klinik und Poliklinik für Psychiatrie und Psychotherapie, München
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kontsekova E, Zilka N, Kovacech B, Skrabana R, Novak M. Identification of structural determinants on tau protein essential for its pathological function: novel therapeutic target for tau immunotherapy in Alzheimer's disease. Alzheimers Res Ther. 2014 Aug 1;6(4):45. doi: 10.1186/alzrt277. eCollection 2014. PMID 25478018
- [Background] Kontsekova E, Zilka N, Kovacech B, Novak P, Novak M. First-in-man tau vaccine targeting structural determinants essential for pathological tau-tau interaction reduces tau oligomerisation and neurofibrillary degeneration in an Alzheimer's disease model. Alzheimers Res Ther. 2014 Aug 1;6(4):44. doi: 10.1186/alzrt278. eCollection 2014. PMID 25478017
- [Background] Novak P, Schmidt R, Kontsekova E, Zilka N, Kovacech B, Skrabana R, Vince-Kazmerova Z, Katina S, Fialova L, Prcina M, Parrak V, Dal-Bianco P, Brunner M, Staffen W, Rainer M, Ondrus M, Ropele S, Smisek M, Sivak R, Winblad B, Novak M. Safety and immunogenicity of the tau vaccine AADvac1 in patients with Alzheimer's disease: a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Neurol. 2017 Feb;16(2):123-134. doi: 10.1016/S1474-4422(16)30331-3. Epub 2016 Dec 10. PMID 27955995